CLINICAL TRIAL: NCT06870032
Title: The Impact of Pulmonary Rehabilitation on Respiratory Function and Quality of Life in Pediatric Patients With Chronic Lung Diseases: A Multidisciplinary Approach in Damietta Governorate
Brief Title: Pulmonary Rehabilitation and Quality of Life in Children With Chronic Lung Diseases: A Multidisciplinary Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Salah El-Sayed, Principal Investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PostDoc_012025
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lung Disease; Quality of Life; Respiratory Function Impaired
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard medical care group (Active Comparator): Patients receiving standard medical care without structured pulmonary rehabilitation.
  Interventions: Other: standard medical care
- structured pulmonary rehabilitation (Other): The experimental group underwent a 12-week structured pulmonary rehabilitation program.
  Interventions: Other: structured pulmonary rehabilitation

INTERVENTIONS:
Other: standard medical care — standard medical care
  Arms: standard medical care group
Other: structured pulmonary rehabilitation — structured pulmonary rehabilitation program including:
  * Physical Therapy: Breathing exercises, airway clearance techniques, inspiratory muscle training.
  * Pediatrics & Chest Medicine: Medical supervision, optimization of pharmacological treatment.
  * Physiology: Monitoring pulmonary function and physiological responses to exercise.
  * Public Health: Evaluating program feasibility and its impact on healthcare utilization.
  Arms: structured pulmonary rehabilitation

SUMMARY:
Chronic lung diseases (CLDs) such as asthma, cystic fibrosis, and bronchopulmonary dysplasia significantly impact pediatric patients' respiratory function and overall well-being. Pulmonary rehabilitation (PR) has been shown to improve lung function, exercise tolerance, and quality of life in affected individuals. However, limited research has been conducted on PR implementation in Egypt.

DETAILED DESCRIPTION:
Pulmonary rehabilitation significantly enhances respiratory function, exercise capacity, and quality of life in pediatric patients with CLDs while reducing healthcare utilization. These findings highlight the necessity of integrating structured PR programs into pediatric respiratory care in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of CLDs, stable clinical condition, and ability to participate in rehabilitation.

Exclusion Criteria:

* Severe comorbidities, recent respiratory infections, or contraindications to physical activity.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in One Second | at basline and after 12-weeks of intervention
  FEV₁ is the volume of air that a person can forcefully exhale in the first second of a forced breath after taking a deep inhalation.
  Interpretation of FEV₁:
  ≥80% of predicted → Normal 60-79% of predicted → Mild obstruction 40-59% of predicted → Moderate obstruction <40% of predicted → Severe obstruction
Forced Vital Capacity | at basline and after 12-weeks of intervention
  FVC is the total volume of air that can be forcefully exhaled after taking the deepest possible breath.
  Normal Values: Typically ≥80% of the predicted value. Obstructive Lung Disease: FVC may be normal or slightly reduced. Restrictive Lung Disease: FVC is significantly reduced due to decreased lung compliance or lung volume.
Peak Expiratory Flow Rate | at basline and after 12-weeks of intervention
  PEFR is the maximum speed of expiration achieved after full lung inflation. It is measured in liters per minute (L/min).
  ormal values depend on age, sex, and height: Adult males: 450-700 L/min Adult females: 300-500 L/min Reduced PEFR: Suggests airway obstruction, such as in asthma or COPD.

SECONDARY OUTCOMES:
Hospitalization Frequency | at basline and after 12-weeks of intervention
  Hospitalization frequency refers to the number of times a patient is admitted to a hospital due to disease exacerbation, complications, or treatment failure.
  Number of hospital admissions within a specific time frame (e.g., per year). Length of hospital stay (days per admission). Emergency department visits requiring inpatient care.
Medication Dependency | at basline and after 12-weeks of intervention
  Medication dependency refers to the extent to which a patient relies on pharmacological treatment to manage symptoms and maintain functional health.
  Frequency and dosage of medication use. Number of rescue medication uses (e.g., bronchodilators in asthma). Reduction or discontinuation of medication over time.
Parental Satisfaction with Treatment | at basline and after 12-weeks of intervention
  Parental satisfaction refers to how parents perceive the effectiveness, convenience, and overall impact of their child's treatment plan.
  Standardized satisfaction surveys (e.g., Likert scale questionnaires). Interviews or focus groups with parents. Feedback on treatment effectiveness, side effects, accessibility, and ease of use.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El-Sayed, Principal Investigator — Horus University in Egypt
Locations (1):
- Out-patient Clinic, Faculty of Physical Therapy, Horus University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided